CLINICAL TRIAL: NCT04859140
Title: Effects of Self-myofascial Release and Manual Massage on Psychometric, Behavioural and Neurophysiological Indexes of Performance and Well-being: a Randomized Control Trial
Brief Title: Selective Effect of Foam Rolling and Manual Massage
Acronym: AUTOMASSEEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Principal Investigator, Prof. Aymeric Guillot, Professor, Laboratoire Interuniversitaire de Biologie de la Motricité
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: LIBMNEURO - AUTOMASSEEG
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Health Behavior; Health, Subjective; Health Knowledge, Attitudes, Practice
Keywords: electroencephalography; electrodermal activity; flexibility; alertness
MeSH Terms: conditions — Health Behavior; Behavior

STUDY DESIGN:
Intervention Model Description: Three independent groups, two measurement points
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation concealment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam rolling (Experimental): The foam rolling routine consisted in unilateral exercises alternatively performed on both legs and bilateral exercises on lower and back muscles. All participants started with the feet in a standing up position with a lacrosse ball. Then, participants performed on the ground the foam rolling exercises with the foam roller targeting leg and back muscles.
  Interventions: Other: Psychometric ratings (Likert-scale); Behavioral: Range of motion measures; Behavioral: Mental calculation task; Device: Resting-state electroencephalography; Device: Resting-state galvanic skin resistance measures
- Manual massage (Experimental): Participants in the manual massage group received manual massage by a professional physiotherapist who was blinded to the purpose of the experiment (20 years of registered practice). Participants were lying in the prone position on a massage table. To facilitate the physiotherapist's maneuvers, massage oil was used. The manual massage protocol reproduced several features of the foam rolling intervention, i.e., order of the areas massaged, massage time per muscles and total duration of the session.
  Interventions: Other: Psychometric ratings (Likert-scale); Behavioral: Range of motion measures; Behavioral: Mental calculation task; Device: Resting-state electroencephalography; Device: Resting-state galvanic skin resistance measures
- Autogenic relaxation (Active Comparator): Participants in the relaxation group listened to a 16 min relaxation audio tape, based on the autogenic training method. Participants were lying on the massage table in supine position, wearing headphones. During this desensitization-relaxation technique, they were guided to visualize bodily perceptions of heaviness and warmth in their arms, thorax and legs. To facilitate concentration, participants were left alone in a dark room.
  Interventions: Other: Psychometric ratings (Likert-scale); Behavioral: Range of motion measures; Behavioral: Mental calculation task; Device: Resting-state electroencephalography; Device: Resting-state galvanic skin resistance measures

INTERVENTIONS:
Other: Psychometric ratings (Likert-scale) — Self-report of perceived anxiety and physical sensations (muscle pain, relaxation and warmth)
Behavioral: Range of motion measures — Sit-and-reach and toe touch tests
Behavioral: Mental calculation task — Iterated substractions (for 2 minutes)
Device: Resting-state electroencephalography — Alpha and beta oscillation power (4 minutes recordings)
Device: Resting-state galvanic skin resistance measures — Skin conductance during the resting state period

SUMMARY:
The present double-blinded randomized controlled design aims at comparing the effects of a full-body manual massage and foam rolling intervention. Sixty-five healthy individuals were randomly allocated to foam rolling, manual massage or a control intervention consisting in an autogenic relaxation routine.

DETAILED DESCRIPTION:
Self-report ratings of perceived anxiety, muscle pain and relaxation were the psychometric outcome variables. Sit-and-reach, toes-touch and mental calculation performances were the behavioral variables. Resting-state alpha and beta power recorded using electroencephalography and galvanic skin resistance measures were the neurophysiological outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Regular practice of foam rolling (10 min routines, 2-3 times per week over the past 6 months)

Exclusion Criteria:

* Chronic medical conditions including functional limitations that might affect proprioception and/or pain perception

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in range of motion measures from standardized flexibility tests | Pretest and an immediate posttest after the intervention
  Lower back and hamstring flexibility index from sit-and-reach and toe touch tests
Resting-state electroencephalography | Pretest and an immediate posttest after the intervention
  Power of alpha and beta neural oscillations
Changes in subjective scores (self-reports on numeric rating scales) | Pretest and an immediate posttest after the intervention
  Perceived anxiety and physical sensations (muscle pain, warmth and relaxation) on a numeric rating scale of 10 cm (0: "Complete absence of anxiety/muscle pain/muscle warmth/muscle relaxation"; 10: "Maximal possible levels of anxiety/muscle pain/muscle warmth/muscle relaxation")
Changes in mental calculation performances | Pretest and an immediate posttest after the intervention
  Iterated substractions for 2 minutes
Changes in physiological arousal | Pretest and an immediate posttest after the intervention
  Skin conductance during resting state periods

CONTACTS AND LOCATIONS:
Locations (1):
- University Claude Bernard Lyon 1, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: Undecided